CLINICAL TRIAL: NCT03453918
Title: Effects of Polyphenols on Iron Absorption in Iron Overload Disorders.
Acronym: POLYFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHU-381; 2017-A01955-48 (Other: 2017-A01955-48)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Dysmetabolic Iron Overload Syndrome; Genetic Hemochromatosis; Iron Absorption; Polyphenols
Keywords: Iron absorption; Polyphenols; Dysmetabolic iron overload syndrome; Metabolic syndrome X; Genetic Hemochromatosis; Oxylipin; Lipidomic analysis
MeSH Terms: conditions — Hemochromatosis; Metabolic Syndrome | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenols (Experimental): patients will receive during the meal, 2 capsules of Oligopin® containing 50 mg of polyphenols each. They will take the two capsules simultaneously with a glass of water, after the starter. Each capsule of Oligopin® contains two excipients: 150 mg of maltodextrin and 30 mg of magnesium stearate.
  Interventions: Dietary Supplement: polyphenols
- Placebo (Experimental): patients will receive during the meal, 2 capsules of placebo, visually identical to Oligopin®. The patient will take the two capsules simultaneously with a glass of water, after the starter. Each capsule of placebo contains two excipients: 218.9 mg of maltodextrin and 1.1 mg of magnesium stearate.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: polyphenols — After 6 hours of fasting, each patient will eat a complete meal course, containing 40 mg of iron, at two different days (wash-out period: 3 days between each meal).
  During each meal, each patient will receive, two capsules containing polyphenols or two placebo capsules (cross-over methodology). The meal in which each patient will receive either polyphenol or placebo will be randomized.
  The diet consists of :
  * Starter: duck gizzard salad.
  * Main course: black pudding and pasta.
  * French cheese.
  * Fruits: kiwi fruit.
  This diet contain approximately 40 mg of iron, with low polyphenol intake. Patients will be asked to eat the whole gizzard and black pudding to ensure the highest iron intake.
  At the end of the meal, blood samples will be collected at 0 minute, 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours, to assess serum iron level, in order to measure the area under the curve of iron kinetic.
  Arms: Polyphenols
Other: Placebo — After 6 hours of fasting, each patient will eat a complete meal course, containing 40 mg of iron, at two different days (wash-out period: 3 days between each meal).
  During each meal, each patient will receive, two capsules containing polyphenols or two placebo capsules (cross-over methodology). The meal in which each patient will receive either polyphenol or placebo will be randomized.
  The diet consists of :
  * Starter: duck gizzard salad.
  * Main course: black pudding and pasta.
  * French cheese.
  * Fruits: kiwi fruit.
  This diet contain approximately 40 mg of iron, with low polyphenol intake. Patients will be asked to eat the whole gizzard and black pudding to ensure the highest iron intake.
  At the end of the meal, blood samples will be collected at 0 minute, 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours, to assess serum iron level, in order to measure the area under the curve of iron kinetic.
  Arms: Placebo

SUMMARY:
Dysmetabolic iron overload syndrome and genetic hemochromatosis are frequent causes of iron overload. Polyphenols are efficient iron-chelators. Investigator hypothesize that polyphenol supplementation can reduce iron absorption in iron overload disease. Iron absorption can be studied by the area-under-the-curve of serum iron after iron oral loading. The primary outcome is the decrease of post-prandial serum iron after rich-iron meal, due to polyphenol supplementation.

DETAILED DESCRIPTION:
Iron overload diseases are highly prevalent. Dysmetabolic iron overload syndrome involves 15% of men with metabolic syndrome X. Genetic hemochromatosis is the most common genetic disease in Northern Europe. Both are due to a lack of regulation in iron absorption. To date, there is no nutritional study for those patients.

Polyphenols, particularly flavanols, have shown as good iron-chelating abilities as pharmacological chelators. However, no human study in iron-overload disease have been so far conducted.

The aim of POLYFER-study is to demonstrate that oral polyphenol intake reduces iron absorption in patients with genetic or metabolic iron-overload diseases.

POLYFER is a cross-over randomized controlled trial comparing the effect of polyphenol supplementation versus placebo on iron absorption after loading dose of iron given through a rich-iron meal. Iron absorption will be studied by the area under the curve of serum iron after the meal. Serum iron will be collected after the meal à 0 minute, 30 minutes, 1 hour, 2 hours, 3 hours et 4 hours.

Because of the nycthemeral variations of serum iron, it is essential to obtain a collection of serum iron data in the basal state (after fasting), allowing the calculation for each subject of a "relative" AUC after iron-rich meal with placebo and after iron-rich meal with polyphenols. The endpoint will be the difference between "relative" AUC after meal rich in iron alone and after polyphenols.

In order to improve the underlying mechanism of atherosclerosis which is highly prevalent in those diseases, we will conduct an ancillary study. Recent studies showed interesting results linking some oxylipins levels and inflammation. Investigator will study basal oxylipin level and post-prandial oxylipin level by lipidomic analysis in both diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Written consent.
* For DIOS Group : at least one criteria of the metabolic syndrome as defined by the International Diabetes Federation, associated with hepatic iron overload measured by MRI (at least 50 µmol/g) or by hepatic biopsy.
* For Genetic Haemochromatosis type 1 Group: homozygosity mutation C282Y in HFE gene ; patients undergoing therapeutic phlebotomies.

Exclusion Criteria:

* Persons under guardianship
* Body-weight less than 45 kg
* Hemoglobin less than 9 g/dL.
* Intestinal malabsorption of any cause
* Current use or previous use during the last 2 months of iron supplement.
* Current use or previous use during the last 2 months of treatment interacting with iron absorption (increasing like C vitamin or decreasing like iron chelators)
* Other causes of hyperferritinemia : chronic inflammatory syndrome, porphyria, hyperferritinemia-cataract-syndrome, chronic alcohol consumption, chronic hemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Decrease of post-prandial iron absorption after dietary polyphenol supplementation | at day 3
  decrease of intestinal iron absorption after standardized oral loading dose through rich-iron meal, expressed by area-under-the-curve of serum iron, due to concomitant administration of a single dose of dietary polyphenos (nutrient complement) versus placebo administration. This outcome is a quantitative variable, treated and analysed as such.

SECONDARY OUTCOMES:
Post-prandial changes of circulating oxylipin in iron overload diseases after iron-rich meal and effects of polyphenols supplementation | at day 1 (fasting versus 3 hours after rich-iron meal, versus 3 hours after rich-iron meal with polyphenol supplementation)
  comparison of oxylipin levels, through lipidomic analyses by spectrophotometry
Comparison of oxylipin levels between DIOS, genetic hemochromatosis and healthy subjects after 6 hours of fasting. | at baseline
  comparison of oxylipin levels, through lipidomic analyses by spectrophotometry. Healthy subjects datas comes from a previous study (MEPHISTO).

CONTACTS AND LOCATIONS:
Overall Officials: Marc RUIVARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Brissot P, Ropert M, Le Lan C, Loreal O. Non-transferrin bound iron: a key role in iron overload and iron toxicity. Biochim Biophys Acta. 2012 Mar;1820(3):403-10. doi: 10.1016/j.bbagen.2011.07.014. Epub 2011 Aug 9. PMID 21855608
- [Background] Gutteridge JM, Rowley DA, Griffiths E, Halliwell B. Low-molecular-weight iron complexes and oxygen radical reactions in idiopathic haemochromatosis. Clin Sci (Lond). 1985 Apr;68(4):463-7. doi: 10.1042/cs0680463. PMID 2578915
- [Background] Brown KE, Dennery PA, Ridnour LA, Fimmel CJ, Kladney RD, Brunt EM, Spitz DR. Effect of iron overload and dietary fat on indices of oxidative stress and hepatic fibrogenesis in rats. Liver Int. 2003 Aug;23(4):232-42. doi: 10.1034/j.1600-0676.2003.00832.x. PMID 12895262
- [Background] Ganz T. Systemic iron homeostasis. Physiol Rev. 2013 Oct;93(4):1721-41. doi: 10.1152/physrev.00008.2013. PMID 24137020
- [Background] Jouanolle AM, Fergelot P, Gandon G, Yaouanq J, Le Gall JY, David V. A candidate gene for hemochromatosis: frequency of the C282Y and H63D mutations. Hum Genet. 1997 Oct;100(5-6):544-7. doi: 10.1007/s004390050549. PMID 9341868
- [Background] Adams PC, Reboussin DM, Barton JC, McLaren CE, Eckfeldt JH, McLaren GD, Dawkins FW, Acton RT, Harris EL, Gordeuk VR, Leiendecker-Foster C, Speechley M, Snively BM, Holup JL, Thomson E, Sholinsky P; Hemochromatosis and Iron Overload Screening (HEIRS) Study Research Investigators. Hemochromatosis and iron-overload screening in a racially diverse population. N Engl J Med. 2005 Apr 28;352(17):1769-78. doi: 10.1056/NEJMoa041534. PMID 15858186
- [Background] Allen KJ, Gurrin LC, Constantine CC, Osborne NJ, Delatycki MB, Nicoll AJ, McLaren CE, Bahlo M, Nisselle AE, Vulpe CD, Anderson GJ, Southey MC, Giles GG, English DR, Hopper JL, Olynyk JK, Powell LW, Gertig DM. Iron-overload-related disease in HFE hereditary hemochromatosis. N Engl J Med. 2008 Jan 17;358(3):221-30. doi: 10.1056/NEJMoa073286. PMID 18199861
- [Background] Mendler MH, Turlin B, Moirand R, Jouanolle AM, Sapey T, Guyader D, Le Gall JY, Brissot P, David V, Deugnier Y. Insulin resistance-associated hepatic iron overload. Gastroenterology. 1999 Nov;117(5):1155-63. doi: 10.1016/s0016-5085(99)70401-4. PMID 10535879
- [Background] Tsuchiya H, Ebata Y, Sakabe T, Hama S, Kogure K, Shiota G. High-fat, high-fructose diet induces hepatic iron overload via a hepcidin-independent mechanism prior to the onset of liver steatosis and insulin resistance in mice. Metabolism. 2013 Jan;62(1):62-9. doi: 10.1016/j.metabol.2012.06.008. Epub 2012 Jul 30. PMID 22854109
- [Background] Le Guenno G, Chanseaume E, Ruivard M, Morio B, Mazur A. Study of iron metabolism disturbances in an animal model of insulin resistance. Diabetes Res Clin Pract. 2007 Sep;77(3):363-70. doi: 10.1016/j.diabres.2007.02.004. Epub 2007 Mar 9. PMID 17350134
- [Background] Ruivard M, Laine F, Ganz T, Olbina G, Westerman M, Nemeth E, Rambeau M, Mazur A, Gerbaud L, Tournilhac V, Abergel A, Philippe P, Deugnier Y, Coudray C. Iron absorption in dysmetabolic iron overload syndrome is decreased and correlates with increased plasma hepcidin. J Hepatol. 2009 Jun;50(6):1219-25. doi: 10.1016/j.jhep.2009.01.029. Epub 2009 Apr 5. PMID 19398238
- [Background] Beaton MD, Chakrabarti S, Levstik M, Speechley M, Marotta P, Adams P. Phase II clinical trial of phlebotomy for non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2013 Apr;37(7):720-9. doi: 10.1111/apt.12255. Epub 2013 Feb 26. PMID 23441892
- [Background] Assi TB, Baz E. Current applications of therapeutic phlebotomy. Blood Transfus. 2014 Jan;12 Suppl 1(Suppl 1):s75-83. doi: 10.2450/2013.0299-12. Epub 2013 Oct 3. No abstract available. PMID 24120605
- [Background] Brune M, Rossander L, Hallberg L. Iron absorption and phenolic compounds: importance of different phenolic structures. Eur J Clin Nutr. 1989 Aug;43(8):547-57. PMID 2598894
- [Background] Hurrell RF, Reddy M, Cook JD. Inhibition of non-haem iron absorption in man by polyphenolic-containing beverages. Br J Nutr. 1999 Apr;81(4):289-95. PMID 10999016
- [Background] Cook JD, Reddy MB, Hurrell RF. The effect of red and white wines on nonheme-iron absorption in humans. Am J Clin Nutr. 1995 Apr;61(4):800-4. doi: 10.1093/ajcn/61.4.800. PMID 7702022
- [Background] Tuntawiroon M, Sritongkul N, Brune M, Rossander-Hulten L, Pleehachinda R, Suwanik R, Hallberg L. Dose-dependent inhibitory effect of phenolic compounds in foods on nonheme-iron absorption in men. Am J Clin Nutr. 1991 Feb;53(2):554-7. doi: 10.1093/ajcn/53.2.554. PMID 1989426
- [Background] Tako E, Beebe SE, Reed S, Hart JJ, Glahn RP. Polyphenolic compounds appear to limit the nutritional benefit of biofortified higher iron black bean (Phaseolus vulgaris L.). Nutr J. 2014 Mar 26;13:28. doi: 10.1186/1475-2891-13-28. PMID 24669764
- [Background] Tako E, Reed SM, Budiman J, Hart JJ, Glahn RP. Higher iron pearl millet (Pennisetum glaucum L.) provides more absorbable iron that is limited by increased polyphenolic content. Nutr J. 2015 Jan 23;14:11. doi: 10.1186/1475-2891-14-11. PMID 25614193
- [Background] Sjodin P, Wallin H, Alexander J, Jagerstad M. Disposition and metabolism of the food mutagen 2-amino-3,8-dimethylimidazo[4,5-f]quinoxaline (MeIQx) in rats. Carcinogenesis. 1989 Jul;10(7):1269-75. doi: 10.1093/carcin/10.7.1269. PMID 2661045
- [Background] Rios-Hoyo A, Cortes MJ, Rios-Ontiveros H, Meaney E, Ceballos G, Gutierrez-Salmean G. Obesity, Metabolic Syndrome, and Dietary Therapeutical Approaches with a Special Focus on Nutraceuticals (Polyphenols): A Mini-Review. Int J Vitam Nutr Res. 2014;84(3-4):113-23. doi: 10.1024/0300-9831/a000198. PMID 26098475
- [Background] Moukette BM, Pieme CA, Njimou JR, Biapa CP, Marco B, Ngogang JY. In vitro antioxidant properties, free radicals scavenging activities of extracts and polyphenol composition of a non-timber forest product used as spice: Monodora myristica. Biol Res. 2015 Mar 14;48(1):15. doi: 10.1186/s40659-015-0003-1. PMID 25885269
- [Background] Tondeur MC, Schauer CS, Christofides AL, Asante KP, Newton S, Serfass RE, Zlotkin SH. Determination of iron absorption from intrinsically labeled microencapsulated ferrous fumarate (sprinkles) in infants with different iron and hematologic status by using a dual-stable-isotope method. Am J Clin Nutr. 2004 Nov;80(5):1436-44. doi: 10.1093/ajcn/80.5.1436. PMID 15531698
- [Background] Ruivard M, Feillet-Coudray C, Rambeau M, Gerbaud L, Mazur A, Rayssiguier Y, Philippe P, Coudray C. Effect of daily versus twice weekly long-term iron supplementation on iron absorption and status in iron-deficient women: a stable isotope study. Clin Biochem. 2006 Jul;39(7):700-7. doi: 10.1016/j.clinbiochem.2006.02.008. Epub 2006 Apr 5. PMID 16603147
- [Background] Hoppe M, Hulthen L, Hallberg L. Serum iron concentration as a tool to measure relative iron absorption from elemental iron powders in man. Scand J Clin Lab Invest. 2003;63(7-8):489-96. doi: 10.1080/00365510310003003. PMID 14743958
- [Background] Andersen SL, Gyrup C, Handberg A, Nielsen GL. Oral iron absorption test should not be performed with iron drops containing ferric iron. Dan Med J. 2015 Aug;62(8):A5116. PMID 26239588
- [Background] Hoppe M, Hulthen L. Validation of the clinical approach of using the induced serum iron increase after 1h as a measure of iron absorption. Clin Nutr. 2006 Feb;25(1):163-5. doi: 10.1016/j.clnu.2005.10.008. Epub 2005 Nov 22. PMID 16307831
- [Background] Kloepfer K, Schmid P, Wuillemin WA, Rufer A. Reference values for oral iron absorption of bivalent iron in healthy volunteers. Swiss Med Wkly. 2015 Jan 22;145:w14063. doi: 10.4414/smw.2015.14063. eCollection 2015. PMID 25612208
- [Background] Kobune M, Miyanishi K, Takada K, Kawano Y, Nagashima H, Kikuchi S, Murase K, Iyama S, Sato T, Sato Y, Takimoto R, Kato J. Establishment of a simple test for iron absorption from the gastrointestinal tract. Int J Hematol. 2011 Jun;93(6):715-719. doi: 10.1007/s12185-011-0878-8. Epub 2011 Jun 1. PMID 21626456
- [Background] Grapov D, Adams SH, Pedersen TL, Garvey WT, Newman JW. Type 2 diabetes associated changes in the plasma non-esterified fatty acids, oxylipins and endocannabinoids. PLoS One. 2012;7(11):e48852. doi: 10.1371/journal.pone.0048852. Epub 2012 Nov 8. PMID 23144998
- [Background] Rametta R, Dongiovanni P, Pelusi S, Francione P, Iuculano F, Borroni V, Fatta E, Castagna A, Girelli D, Fargion S, Valenti L. Hepcidin resistance in dysmetabolic iron overload. Liver Int. 2016 Oct;36(10):1540-8. doi: 10.1111/liv.13124. Epub 2016 Apr 6. PMID 26998752
- [Background] Gladine C, Newman JW, Durand T, Pedersen TL, Galano JM, Demougeot C, Berdeaux O, Pujos-Guillot E, Mazur A, Comte B. Lipid profiling following intake of the omega 3 fatty acid DHA identifies the peroxidized metabolites F4-neuroprostanes as the best predictors of atherosclerosis prevention. PLoS One. 2014 Feb 18;9(2):e89393. doi: 10.1371/journal.pone.0089393. eCollection 2014. PMID 24558496
- [Background] Kim J, Carlson ME, Kuchel GA, Newman JW, Watkins BA. Dietary DHA reduces downstream endocannabinoid and inflammatory gene expression and epididymal fat mass while improving aspects of glucose use in muscle in C57BL/6J mice. Int J Obes (Lond). 2016 Jan;40(1):129-37. doi: 10.1038/ijo.2015.135. Epub 2015 Jul 29. PMID 26219414
- [Background] Gouveia-Figueira S, Spath J, Zivkovic AM, Nording ML. Profiling the Oxylipin and Endocannabinoid Metabolome by UPLC-ESI-MS/MS in Human Plasma to Monitor Postprandial Inflammation. PLoS One. 2015 Jul 17;10(7):e0132042. doi: 10.1371/journal.pone.0132042. eCollection 2015. PMID 26186333
- [Background] Lobbes H, Gladine C, Mazur A, Pereira B, Duale C, Cardot JM, Ruivard M. Effect of procyanidin on dietary iron absorption in hereditary hemochromatosis and in dysmetabolic iron overload syndrome: A crossover double-blind randomized controlled trial. Clin Nutr. 2020 Jan;39(1):97-103. doi: 10.1016/j.clnu.2019.02.012. Epub 2019 Feb 11. PMID 30792142